CLINICAL TRIAL: NCT01322815
Title: A Pilot Trial of GI-4000 Plus Bevacizumab and Either FOLFOX or FOLFIRI in Patients With Ras Mutant Positive Metastatic Colorectal Cancer, Either Newly Diagnosed or Previously Treated.
Brief Title: A Pilot Trial of GI-4000 Plus Bevacizumab and Either FOLFOX or FOLFIRI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual rate
Sponsor: Georgetown University (Other)
Collaborators: GlobeImmune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI-4000-05
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-02

CONDITIONS: Colon Cancer
Keywords: colon cancer; metastatic; vaccine
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis | interventions — Drug Therapy; Fluorouracil; Leucovorin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy and GI-4000 (Experimental): Standard chemotherapy and bevacizumab 40 yeast units (YU) GI-4000 prior to initiation of chemotherapy and then intercycle 7 days after each chemotherapy cycle for up to 8 cycles.
  maintenance of GI-4000 injection and bevacizumab every 2 weeks
  Interventions: Drug: chemotherapy and GI-4000
- GI-4000 and bevacizumab (Experimental): maintenance with GI-4000 and bevacizumab for patients who have completed first-line chemotherapy
  Interventions: Drug: GI-4000

INTERVENTIONS:
Drug: chemotherapy and GI-4000 — Standard chemotherapy and bevacizumab 40YU GI-4000 prior to initiation of chemotherapy and then intercycle 7 days after each chemotherapy cycle for up to 8 cycles.
  maintenance of GI-4000 injection and bevacizumab every 2 weeks
  Other Names: 5-fluorouracil (5-FU), leucovorin. oxaliplatin; 5-fluorouracil (5-FU), leucovorin, irinotecan; avastin
  Arms: Chemotherapy and GI-4000
Drug: GI-4000 — 40 YU GI-4000 every 2 weeks Bevacizumab every 2 weeks
  Other Names: Avastin
  Arms: GI-4000 and bevacizumab

SUMMARY:
The purpose of this study is to test the safety of GI-4000 and see what effects (good and bad) it has against cancer over time. This study is also being done to measure the immune response to GI-4000. Study drug will be given in addition to a standard of care which is a standard therapy given to patients with your type of cancer (colon).

DETAILED DESCRIPTION:
Subject visits will occur 1-4 weeks prior to initiation of GI-4000, then

* In newly diagnosed (Group A) patients, at every FOLFOX/FOLFIRI plus bevacizumab visit, bevacizumab and GI-4000 dosing visit, GI-4000 dosing visit and then quarterly after completion of therapy
* In patients with stable disease who have completed a first line therapy with an oxaliplatin or irinotecan plus fluoropyrimidine and bevacizumab containing regimen (Group B), at every bevacizumab and GI-4000 dosing visit, GI-4000 dosing visit and then quarterly after completion of therapy

Group A patients (N=26) will be enrolled into the study prior to the initiation of first line therapy with bevacizumab plus either FOLFOX (N=13) or FOLFIRI (N=13)

* Subjects will receive 1 40 yeast units (YU) dose of GI-4000 prior to initiation of FOLFOX or FOLFIRI plus bevacizumab, then intercycle doses of GI-4000 will be given 7 days after each cycle while first line therapy is given (up to 8 cycles)
* After completion of first line therapy, subjects will enter the maintenance phase in which bevacizumab and GI-4000 will be given concurrently every 2 weeks for as long as therapy can be tolerated or until progression
* If a subject discontinues bevacizumab therapy due to intolerance, the subject will continue GI-4000 every 2 weeks until progression, intolerance or withdrawal from the study

Group B patients (N=26) with stable disease who have completed a first line therapy with an oxaliplatin or irinotecan plus fluoropyrimidine and bevacizumab containing regimen ) will enter the trial prior to receiving therapy with bevacizumab

* Subjects will receive 40 yeast unit (YU) GI-4000 concurrently with each bevacizumab dose for as long as therapy can be tolerated or until progression
* If a subject discontinues bevacizumab therapy due to intolerance, the subject will continue GI-4000 every 2 weeks until progression, intolerance or withdrawal from the study

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic colorectal cancer with a Ras mutation
* Measurable or evaluable disease
* No prior therapy fore metastatic disease except for group A: > 6 months since completion of adjuvant therapy and Group B: those patients who enroll just after completing bevacizumab plus FOLFOX or FOLFIRI
* Anticipated survival of at least 6 months
* Ambulatory with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Ability to maintain weight
* Normal organ and marrow function
* Women of child-bearing potential and men must agree to avoid pregnancy or fathering a child for the duration of study participation and for 6 months after the final scheduled study visit.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Prior chemotherapy other than that listed in inclusion criteria
* Receiving any other investigational agent
* Known brain metastases, uncontrolled seizure disorders, encephalitis, or multiple sclerosis
* History of known hypersensitivity to S. cerevisiae, bevacizumab or any component of FOLFOX or FOLFIRI
* Concurrent and chronic therapy with corticosteroids or any other immunosuppressive drugs
* Uncontrolled hypertension, unstable angina, congestive heart failure, peripheral vascular disease, serious cardiac arrythmias requiring medication
* History of heart attack or stroke within 6 months before enrollment
* History of intra-abdominal abscess, abdominal fistula, gastrointestinal perforation, or active peptic ulcer disease
* Bleeding disorder or coagulopathy
* Serious non-healing wound, ulcer or bone fracture
* Major surgical procedure, open biopsy, or traumatic injury within 4 weeks prior to enrollment or anticipation of need for surgery during the study
* Known active infection with HIV, hepatitis B or C
* History of splenectomy
* History of Crohn's disease or ulcerative colitis
* History of organ transplantation
* Evidence of immunodeficiency or immune suppression
* Any Autoimmune disease
* Active infection
* Concurrent malignancy
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Marshall, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy and GI-4000: Standard chemotherapy and bevacizumab 40YU GI-4000 prior to initiation of chemotherapy and then intercycle 7 days after each chemotherapy cycle for up to 8 cycles.
  maintenance of GI-4000 injection and bevacizumab every 2 weeks
  chemotherapy and GI-4000: Standard chemotherapy and bevacizumab 40YU GI-4000 prior to initiation of chemotherapy and then intercycle 7 days after each chemotherapy cycle for up to 8 cycles.
  maintenance of GI-4000 injection and bevacizumab every 2 weeks
Period: Overall Study
Arm/Group | Chemotherapy and GI-4000 | GI-4000 and Bevacizumab
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with RAS mutant positive metastatic colorectal cancer (CRC), either having received prior 1st-line therapy with an oxaliplatin or irinotecan plus fluoropyrimidine and bevacizumab containing regimen, or no prior therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy and GI-4000 | GI-4000 and Bevacizumab | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 48 [35 to 71] | 45 [42 to 51] | 45 [35 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11
Prior treatment status [Number; unit: participants]
  Prior 1st-line therapy | 0 | 4 | 4
  No prior therapy | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Alive and Free of Progression at 4 Months (Patients Who Have Undergone Prior Therapy) and 10 Months (Untreated Patients)
Description: Clinical benefit rate is defined as the proportion of patients alive and free of progression at 4 Months (Patients Who Have Undergone Prior Therapy) and 10 Months (Untreated Patients), assessed from first treatment with GI-4000. Progression is defined as CR (complete response) = disappearance of all target lesions; PR (partial response) = 30% decrease in the sum of the longest diameter of the target lesions; PD (progressive disease) = 20% increase in the sum of the longest diameter of the target lesions; or SD (stable disease) = small changes that do not meet the above criteria.
Time Frame: 4 Months for patients who had undergone prior 1st-line therapy, and 10 months for previously untreated patients
Population: Patients with RAS mutant positive metastatic colorectal cancer (CRC), either newly diagnosed, or having completed first line therapy with an oxaliplatin or irinotecan plus fluoropyrimidine and bevacizumab containing regimen.
Measure: Number; unit: participants
Arm/Group | Chemotherapy and GI-4000 | GI-4000 and Bevacizumab
Number analyzed (Participants) | 7 | 4
participants | 4 | 2

ADVERSE EVENTS:
Time Frame: From 48 to 739 days: as long as each individual patient was on study (from Nov 2010 until Sep 2013)
Arm/Group | Chemotherapy and GI-4000 | GI-4000 and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/4
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy and GI-4000 (N=7) | GI-4000 and Bevacizumab (N=4)
thrombosis (Cardiac disorders) | 1 (1) | 0 (0) — Unlikely related to GI-4000. Probably related to chemotherapy.
low neutrophil count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Unlikely related to GI-4000. Probably related to chemotherapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy and GI-4000 (N=7) | GI-4000 and Bevacizumab (N=4)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Fatigue (General disorders) | 4 (5) | 1 (1)
flu (General disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 1 (1)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Vaginismus (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No